CLINICAL TRIAL: NCT00864916
Title: A Randomized, Placebo-Controlled Trial of Pentoxifylline Plus Combination ART vs. Combination ART Alone to Improve Endothelial Dysfunction in HIV-Infected Patients
Brief Title: Pentoxifylline and Combination Antiretroviral Therapy to Improve Blood Vessel Function in HIV-Infected People
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Samir K Gupta, MD, MS, Associate Professor of Medicine, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 646; R01HL095149 (NIH)
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-04

CONDITIONS: HIV; Vascular Diseases; Cardiovascular Diseases; Atherosclerosis; HIV Infections
Keywords: Endothelial Function; Pentoxifylline; Antiretroviral Therapy; Inflammation
MeSH Terms: conditions — Vascular Diseases; Cardiovascular Diseases; Atherosclerosis; HIV Infections; Inflammation | interventions — Antiretroviral Therapy, Highly Active; Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive pentoxifylline and combination antiretroviral therapy (cART).
  Interventions: Drug: Combination antiretroviral therapy (cART); Drug: Pentoxifylline
- 2 (Active Comparator): Participants will receive placebo and cART.
  Interventions: Drug: Combination antiretroviral therapy (cART); Drug: Placebo

INTERVENTIONS:
Drug: Combination antiretroviral therapy (cART) — Participants will receive the appropriate cART medications, as prescribed by their primary HIV doctor for 48 weeks. (cART medications may be prescribed beyond the length of this study.)
Drug: Pentoxifylline — Participants will receive 400 mg of pentoxifylline three times per day for 48 weeks.
  Arms: 1
Drug: Placebo — Participants will receive placebo three times per day for 48 weeks.
  Arms: 2

SUMMARY:
People infected with HIV have a greater risk of developing cardiovascular disease than people not infected with HIV. This may be due to increased inflammation in the blood vessels. This study will determine whether an anti-inflammatory drug, pentoxifylline, in combination with antiretroviral medications, is more effective at improving blood vessel function and reducing inflammation than antiretroviral medications alone in people infected with HIV.

DETAILED DESCRIPTION:
People infected with HIV have an increased risk for cardiovascular disease, which is a leading cause of death for those with HIV. This may be due to increased inflammation of the blood vessels, which is often observed in HIV-infected people and which can lead to endothelial dysfunction-a condition that involves the malfunctioning of the thin layer of cells that line the interior surface of blood vessels. Endothelial dysfunction increases the risk of developing both atherosclerosis and cardiovascular disease.

Much of the focus on the causes of HIV-related endothelial dysfunction has been centered on the use of several types of antiretroviral medications used to treat HIV infection. However, more recent data suggest that newer protease inhibitors, a type of antiretroviral medication, are not associated with endothelial dysfunction and that newer combination antiretroviral therapy (cART) regimens result in an initial improvement in endothelial dysfunction. Yet, preliminary research has also shown that in people who receive cART, the risk of endothelial dysfunction in fact persists with time, suggesting that a mechanism other than viral control, notably inflammation, is playing a role in endothelial dysfunction. Pentoxifylline is a medication that is currently used to reduce leg pain in people with blockages in the blood vessels in their legs. Previous research has shown that pentoxifylline may improve blood vessel function and reduce inflammation in people infected with HIV, but more research is needed to confirm these benefits. The purpose of this study is to compare the safety and effectiveness of pentoxifylline and cART versus cART alone at improving endothelial function and reducing inflammation in HIV-infected people.

This study will enroll people infected with HIV who are about to start receiving cART. At a baseline study visit, participants will undergo a medical history review; physical examination; measurements of blood pressure, heart rate, height, weight, temperature, waist, and hip; and blood and urine collection. An ultrasound imaging test of the arm will measure blood vessel function. Participants will then be randomly assigned to receive either pentoxifylline or placebo three times a day for 48 weeks. All participants will also receive cART medications, as prescribed by their primary HIV doctor. At study visits at Weeks 4, 8, 16, 24, 32, and 48, participants will undergo repeat baseline measurements; however, the ultrasound testing will only occur at Weeks 8, 24, and 48.

ELIGIBILITY:
Inclusion Criteria:

* Documentation of HIV infection with a positive HIV enzyme-linked immunosorbent assay (ELISA) test and confirmatory western blot test
* Has not received any antiretroviral therapies in the 6 months before screening
* Participant is planning to initiate cART, per the primary HIV caregiver (there is no CD4 or HIV-1 RNA level criteria)

Exclusion Criteria:

* Incarceration at the time of screening or at any study visit
* Diagnosed vascular disease, including history of angina pectoris, coronary disease, peripheral vascular disease, cerebrovascular disease, aortic aneurysm, or otherwise known atherosclerotic disease
* Diagnosed disease or process, other than HIV infection, associated with increased systemic inflammation (including, but not limited to, systemic lupus erythematosis, inflammatory bowel diseases, or other collagen vascular diseases). Hepatitis B or C co-infections are NOT exclusionary.
* History of bleeding diathesis, gastrointestinal ulceration or bleeding, cerebrovascular aneurysm or bleeding, or retinal hemorrhage
* Known or suspected cancer requiring systemic treatment in the 6 months before screening
* History of American Diabetes Association (ADA)-defined diabetes mellitus. History of gestational diabetes is not exclusionary.
* History of migraine headaches
* History of Raynaud's phenomenon
* History of cardiac arrhythmias or cardiomyopathy
* History of hypothyroidism or hyperthyroidism, even if treated
* Known allergy or intolerance to pentoxifylline or other methylxanthines (e.g., theophylline, caffeine, theobromine). Use of caffeinated products, except on the mornings of the study visits, is not exclusionary.
* Known allergy or intolerance to nitroglycerin
* History of carotid bruits
* Creatinine clearance less than 50 mL/min, using the Cockcroft-Gault equation and a serum creatinine level measured in the 28 days before screening or at the screening visit
* Hemoglobin less than 9.0 mg/dL in the 28 days before screening or at the screening visit
* Alanine aminotransferase (ALT) level or aspartate aminotransferase (AST) greater than three times the upper limit of normal (ULN) in the 28 days before screening or at the screening visit
* Total bilirubin greater than 2.5 times ULN in the 28 days before screening or at the screening visit
* Fever, defined as a temperature greater than or equal to 38.0 degrees Celsius (C) in the 48 hours before screening. Fever in the 48 hours before each study visit will require postponement of that study visit until the participant's temperature has been lower than 38.0 C for at least 48 hours; fevers continuing past the allowed study visit timeframe will result in study discontinuation.
* Therapy for acute infection or other serious medical illnesses (besides HIV infection) within 14 days prior to screening.

Note: Therapy for acute infection or other serious medical illnesses that overlaps with a main study visit will result in postponement of that study visit until the course of therapy is completed; postponement outside of the allowed study visit timeframe will result in study discontinuation.

* Pregnancy or breastfeeding during the course of the study.
* Hypotension, defined as systolic blood pressure < 90mmHg, at time of screening.

Note: Hypotension noted prior to brachial artery reactivity testing on each main study visit will result in study visit postponement of at least one day until systolic pressure is ≥ 90mmHg the morning of brachial reactivity testing; postponement outside of the allowed study visit timeframe will result in study discontinuation.

* Uncontrolled hypertension, defined as a confirmed systolic blood pressure > 160mmHg at screening (regardless of use of antihypertensive medications).
* Receipt of anti-inflammatory agents (including, but not limited to, plaquenil, infliximab, etanercept, mycophenylate mofetil, sirolimus, tacrolimus, cyclosporine, pentoxifylline, thalidomide).
* Receipt of investigational agents, cytotoxic chemotherapy, systemic or topical glucocorticoids (of any dose), or anabolic steroids within 28 days of screening.

Note: Physiologic testosterone replacement therapy is not exclusionary.

* Receipt of lipid-lowering drugs, acetazolamide, anticoagulants, anticonvulsants, or thyroid replacements within 28 days prior to screening.
* Receipt of aspirin or other NSAIDS within 7 days of screening.
* Use of sildenafil, vardenafil, or tadalafil within 72 hours (before or after) of each main study visit.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-03; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir K. Gupta, MD, MS, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Infectious Diseases Research Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PTX+cART: Participants will receive pentoxifylline and combination antiretroviral therapy (cART).
  Combination antiretroviral therapy (cART): Participants will receive the appropriate cART medications, as prescribed by their primary HIV doctor for 48 weeks. (cART medications may be prescribed beyond the length of this study.)
  Pentoxifylline: Participants will receive 400 mg of pentoxifylline three times per day for 48 weeks.
- Placebo+cART: Participants will receive placebo and cART.
  Combination antiretroviral therapy (cART): Participants will receive the appropriate cART medications, as prescribed by their primary HIV doctor for 48 weeks. (cART medications may be prescribed beyond the length of this study.)
  Placebo: Participants will receive placebo three times per day for 48 weeks.
Period: Overall Study
Arm/Group | PTX+cART | Placebo+cART
Started | 10 | 9
Completed | 4 | 5
Not Completed | 6 | 4
Not completed — Lost to Follow-up | 4 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Completed enrollment visit
Groups:
- Total: Total of all reporting groups
Arm/Group | PTX+cART | Placebo+cART | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (12.1) | 34.0 (8.8) | 36.0 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 9 | 7 | 16
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Flow-mediated Dilation of the Brachial Artery
Description: Flow-mediated dilation (% dilation of the brachial artery) at week 48
Time Frame: Measured at Week 48
Population: Numbers of participants who completed the week 48 visit procedures
Measure: Mean (Standard Deviation); unit: percent dilation of the brachial artery
Arm/Group | PTX+cART | Placebo+cART
Number analyzed (Participants) | 4 | 5
percent dilation of the brachial artery | 2.25 (2.92) | 3.36 (1.44)
Statistical Analysis 1: Comparison: PTX+cART vs Placebo+cART; Test type: Superiority or Other; p = 0.52, Regression, Linear; Mean Difference (Final Values) = -1.34

ADVERSE EVENTS:
Arm/Group | PTX+cART | Placebo+cART
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 6/10 | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PTX+cART (N=10) | Placebo+cART (N=9)
Gastrointestinal upset (Gastrointestinal disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No